CLINICAL TRIAL: NCT05410158
Title: Comparative Study of Ketamine Added to Bupivacaine in PECS Block Versus Topical Wound Instillation on Post Operative Analgesia in Modified Radical Mastectomy Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saif Eldeen Gamal Khalaf, Comparative study of ketamine added to bupivacaine in PECS block versus topical wound instillation on post operative analgesia in modified radical mastectomy surgery, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ketamine analgesic efficacy
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-03

CONDITIONS: Ketamine, Pecs Block, Topical Wound Instillation , Modefied Radical Mastectomy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecs block group (Other): The Pecs block will be performed while the patient in the supine position with the ipsilateral upper limb abducted 90 degree with an 80 mm 21 G needle (Pajunk®SonoPlex Stim cannula U.S.A) using linear array ultrasound probe of high frequency (Sonosite®, Inc. U.S.A) starting from the lateral third of the clavicle and moving distally and laterally to the mid axillary line .
  Patients will be given ultrasound guided, modified Pecs block with 30 mL of 0.25% bupivacaine hydrochloride (Markyrene ®Sigma Tec, Egypt) plus ketamine hydrochloride (1 mg/kg) (Ketamine® Sigma-Tec, Egypt) injected between the pectoralis minor and the serratus anterior muscles , and skin incision will be performed 15 minutes after the block was given.
  Interventions: Drug: Ketamine in PECS block versus topical wound instillation
- Topical instillation group: (Other): After surgical hemostasis before wound closure Patients will receive 1 mg/kg ketamine hydrochloride plus 30 mL of 0.25% bupivacaine hydrochloride which will be put in asterile syringe and irrigated onto the surgical field at the end of surgery .
  Interventions: Drug: Ketamine in PECS block versus topical wound instillation

INTERVENTIONS:
Drug: Ketamine in PECS block versus topical wound instillation — On arrival to the operating room, an intravenous line will be inserted in the contralateral upper limb to the side of surgery. Anesthesia will be induced for all participating patients with 2 μg/kg fentanyl, 2 - 3 mg/kg propofol and 1.5 mg/kg lidocaine. Endotracheal intubation will be facilitated by 0.15 mg/kg cis-atracurium.The patients will be randomly assigned into 2 groups ( pecs block group , topical instillation group) using a randomization-computer program . Anesthesia will be maintained by 1 - 1.5 MAC isoflurane in 50% oxygen/ air mixture and 0.03 mg/kg cisatrcurium, respectively, in ventilation parameters that maintain normocapnia. At the end of surgery, a reversal of the muscle relaxant will be done using neostigmine (0.04 mg/kg) and atropine (0.01 mg/kg). After extubation, all patients will be transmitted to the post anesthesia care unit (PACU) for follow up .

SUMMARY:
Comparative study of ketamine added to bupivacaine in PECS block versus topical wound instillation on post operative analgesia in modified radical mastectomy surgery

ELIGIBILITY:
Inclusion Criteria:

- 1) female patients aged 18 - 60 years, 2) American Society of Anesthesiologists (ASA) class | , || , ||| 3) With body weight of 50 - 90 kg . 4) female patients diagnosed with cancer breast and scheduled for modified radical mastectomy .

5) patients not known to be allergic to any of the medications used in the study.

Exclusion Criteria:

- 1) patients with known allergy to the study drugs . 2) patients with significant cardiac, respiratory, renal or hepatic disease . 3) patients with drug or alcohol abuse . 4) patients with psychiatric illness that would interfere with perception and assessment of pain.

5) Patients with a history of bleeding diathesis; opioid dependence; sepsis; prior surgery in the supraclavicular, infraclavicular or axillary regions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-07-28 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
- The primary outcome measure in this study will be the total dose of morphine consumption during the 48 hours Postoperatively. | july 2022 - feb 2023